CLINICAL TRIAL: NCT03431441
Title: Clinical Evaluation of 2-Week Reusable ACUVUE 2 Vivid Style
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6180
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Visual Acuity

STUDY DESIGN:
Masking Description: Due to visible print differences, subjects and investigators will be aware of the patterns/variants of the investigational product. However, subjects will be masked to the lens brand to prevent bias during the lens discussions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- JJVC Marketed Contact Lens (Experimental): ACUVUE 2 Vivid Style
  Interventions: Device: JJVC Marketed Contact Lens

INTERVENTIONS:
Device: JJVC Marketed Contact Lens — Female subjects that are habitual contact lens wearers between the ages of 18 to 39 will be dispensed 1 treatment of the JJVC Marketed Contact Lens during the 2-visit study.

SUMMARY:
This will be a single site, non-randomized, dispensing, brand-masked to the subject, bilateral single treatment study. There will be 2 study visits with a 10 to 14-day contact lens wear period between visits.

ELIGIBILITY:
Inclusion Criteria:

-Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol (i.e., willing to wear only the study lenses and not use habitual lenses during the study).
3. Females between 18 and 39 (inclusive) years of age at the time of screening.
4. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye.
5. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye.
6. Have spherical best corrected visual acuity of 20/30 or better in each eye.
7. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report.
8. The subject must be willing to be photographed and/or video-taped.

Exclusion Criteria:

1. Currently pregnant or lactating
2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion).
3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion).
4. Any previous, or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.).
5. Any previous history or signs of a contact lens-related corneal inflammatory event (eg, past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear.
6. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment.
7. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician).

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VRC East, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 subjects were enrolled in the study. Of those enrolled, 24 subjects were assigned and administered. Of the total assigned subjects, 19 subjects completed the study, while 5 subjects were discontinued from the study.
Groups:
- Test: Subject that wore the etafilcon A lenses throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Test
Started (24) | 24
Completed (19) | 19
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2
Not completed — Dispensed Incorrect Replacement Lens | 1

BASELINE CHARACTERISTICS:
Arm/Group | Test
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Year] | 28.6 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: LogMAR Objective Vision (High Illumination/High Contrast)
Description: Monocular high illuminance high contrast VA with the study lenses was collected to the nearest letter using computer generated logMAR charts. 0.02 logMAR is equivalent to 1 letter. Negative logMAR values indicate better lens performance. The average visual acuity was reported for each lens type.
Time Frame: 5 minutes after lens fitting
Population: All subjects who received at least one study article regardless of the randomization status.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Test
Number analyzed (Participants) | 24
Number analyzed (Eyes) | 46
logMAR | -0.105 (0.0546)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study, approximately 10 to 14 days per subject.
Arm/Group | Test
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT03431441/Prot_SAP_000.pdf